CLINICAL TRIAL: NCT00718406
Title: Pain Relief of Metoprolol Versus Metoprolol Plus Morphine in Acute Chest Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Other Study IDs: S203-02
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2002-08

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute coronary syndrome; Chest pain; Betablockers; Morphine; Prehospital phase
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain | interventions — Metoprolol; Morphine

ARMS (2):
- A (Active Comparator): A=metoprolol
  Interventions: Drug: Metoprolol
- B (Active Comparator): B=metoprolol plus morphine
  Interventions: Drug: metoprolol plus morphine

INTERVENTIONS:
Drug: Metoprolol
  Arms: A
Drug: metoprolol plus morphine
  Arms: B

SUMMARY:
The primary aim was to evaluate the relief of chest pain during the first 30 minutes among patients who received metoprolol alone as compared with metoprolol plus morphine

ELIGIBILITY:
Inclusion Criteria:

* Acute chest pain
* ECG-signs indicating myocardial ischemia

Exclusion Criteria:

* Heart rate < 60 beats/min
* Systolic blood pressure < 110 mmHg
* High degree AV-block
* Signs of obstructive pulmonary disease
* Signs of pulmonary oedema
* Unwillingness
* Participation in other studies
* Long delay between arrival of ambulance and randomisation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Institution, Dept of Molecular and Clinical Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden